CLINICAL TRIAL: NCT02780700
Title: LUME-Colon 2: An Open-label Randomized Phase II Study to Assess the Efficacy and Safety of Nintedanib Alone or in Combination With Capecitabine for Patients With Refractory Metastatic Colorectal Cancer
Brief Title: Nintedanib Alone or in Combination With Capecitabine in Refractory Metastatic Colorectal Cancer [LUME-Colon 2]
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Substance discontinued
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199.251
Record Dates: First submitted 2016-05-20; First posted 2016-05-23 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — nintedanib; Capecitabine

ARMS (2):
- Nintedanib (Experimental)
  Interventions: Drug: Nintedanib
- Nintedanib plus capecitabine (Experimental)
  Interventions: Drug: Nintedanib; Drug: Capecitabine

INTERVENTIONS:
Drug: Nintedanib
Drug: Capecitabine
  Arms: Nintedanib plus capecitabine

SUMMARY:
The objective of this Phase II study is to assess the efficacy and safety of nintedanib alone or in combination with capecitabine for patients with refractory metastatic colorectal cancer (mCRC) after failure of at least 2 lines of standard treatment

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed colorectal adenocarcinoma
* Metastatic or locally advanced disease not amenable to curative surgery and/or radiotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status <= 1
* At least one measurable lesion according to RECIST 1.1
* Previously treated with all of the following: fluoropyrimidine, (e.g. 5-fluorouracil (5-FU), capecitabine or TAS-102); oxaliplatin: Patients treated with oxaliplatin in adjuvant setting should have progressed within 6 months of completion of adjuvant therapy or they must have been treated with oxaliplatin for metastatic disease; Irinotecan; Vascular Endothelial Growth Factor (VEGF) directed treatment (e.g. bevacizumab, aflibercept, ramucirumab or regorafenib); cetuximab or panitumumab for patients with K-Ras wt or Ras wt tumors
* Minimal time interval of 3 weeks between the last administration of Colorectal Cancer (CRC) treatment (cytotoxics or targeted agents) and starting of trial therapy
* Adequate liver and kidney function
* Further inclusion criteria apply

Exclusion criteria:

* Prior treatment with nintedanib.
* Any other investigational agent received within 3 weeks prior to randomization
* Known hypersensitivity or intolerability to the trial drugs or their excipients
* History of other malignancies in the last 5 years, in particular those that could interfere with interpretation of results. Patients with adequately treated basal or squamous cell skin cancer or cervix carcinoma and other early stage cancer treated curatively are eligible
* History of severe or unexpected reactions to fluoropyrimidine therapy or any of its excipients
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Treatment with sorivudine or its chemically related analogues, such as brivudine
* Serious concomitant disease or medical condition affecting compliance with trial requirements or which are considered relevant for the evaluation of the efficacy or safety of the trial drug, such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with trial participation or trial drug administration, and in the judgment of the investigator would make the patient inappropriate for entry into the trial
* Major injuries and/or surgery or bone fracture within 4 weeks of trial inclusion (signing Informed Consent), or planned surgical procedures during the trial period
* Significant cardiovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of myocardial infarction within past 6 months of trial inclusion, congestive heart failure > New York Heart Association (NYHA) II)
* History of severe hemorrhagic or thromboembolic event in the past 6 months (excluding central venous catheter thrombosis and peripheral deep vein thrombosis). Known inherited predisposition to bleeding or to thrombosis
* Bleeding or thrombotic disorders requiring anticoagulant therapy such as warfarin, or similar agents requiring therapeuticInternational normalized ratio (INR) monitoring (treatment with low molecular weight heparin and/or heparin flush as needed for maintenance of an indwelling intravenous device is allowed)
* Inflammatory bowel disease and other serious medical conditions increasing the risk of perforation or bleeding according to investigator's judgment
* Gastrointestinal disorders or abnormalities that would interfere with absorption of study drug
* Patient with brain metastases that are symptomatic and/or require therapy. Patients with previously treated and stable brain metastases are allowed
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-07-05; Primary Completion 2016-09-09 (Actual); Study Completion 2016-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Fort Wayne Medical Oncology Hematology, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an exploratory, phase II multi-center, non-comparative, open-label, randomized trial to assess the efficacy and safety of nintedanib alone, or in combination with capecitabine in patients with refractory metastatic colorectal cancer.
Pre-assignment Details: Patients eligible for this study were to be randomized in a 1:1 fashion to receive either nintedanib alone or combination with capecitabine.
  One patient with combination therapy entered study, no patient with nintedanib alone entered study.
Groups:
- Nintedanib Plus Capecitabine: Patients were to be orally administered tablets of Nintedanib and 1000 mg/m2 Capecitabine twice daily.
  Nintedanib: 21 day cycles; Capecitabine: first 14 days of each 21 day cycle
Period: Overall Study
Arm/Group | Nintedanib Plus Capecitabine
Started | 1
Completed | 0
Not Completed | 1
Not completed — Progressive disease | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This will comprise all patients who are randomized and are documented to have taken at least one dose of trial medication
Arm/Group | Nintedanib Plus Capecitabine
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: TS
  years | 50 (NA) — Not Applicable as only one patient was treated
Sex: Female, Male [Count of Participants; unit: Participants] — Population: TS
  Participants
    Female | 1
    Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: TS
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 0
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: TS
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 1
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization until objective tumor progression or death.
  Since only one patient was enrolled prior to termination of the trial, no data summarization or analysis was carried out.
Time Frame: Data collected up to cut-off date 09 Sep 2016, Up to 02 months
Population: Randomized set (RS): Comprising all patients who have a randomization date recorded in the electronic Case record form (eCRF).
Measure: Median (Full Range); unit: months
Arm/Group | Nintedanib Plus Capecitabine
Number analyzed (Participants) | 1
months | NA [NA to NA] — Since only one patient was enrolled prior to termination of the trial, no data summarization or analysis was carried out.

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization until death from any cause.
  Since only one patient was enrolled prior to termination of the trial, no data summarization or analysis was carried out.
Time Frame: Data collected up to cut-off date 09 Sep 2016, Up to 02 months
Population: RS
Measure: Median (Full Range); unit: months
Arm/Group | Nintedanib Plus Capecitabine
Number analyzed (Participants) | 1
months | NA [NA to NA] — Since only one patient was enrolled prior to termination of the trial, no data summarization or analysis was carried out.

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
  Since only one patient was enrolled prior to termination of the trial, no data summarization or analysis was carried out.
Time Frame: tumor response was to be assessed by imaging according to RECIST (version 1.1) every 6 weeks.
Population: RS
Measure: Number; unit: Percentage of participants
Arm/Group | Nintedanib Plus Capecitabine
Number analyzed (Participants) | 1
Percentage of participants | NA — Since only one patient was enrolled prior to termination of the trial, no data summarization or analysis was carried out.

4. Secondary Outcome: Disease Control (DC)
Description: Disease control is defined as CR or PR or Stable disease (SD) per RECIST version 1.1.
  Since only one patient was enrolled prior to termination of the trial, no data summarization or analysis was carried out.
Time Frame: Data collected up to cut-off date 09 Sep 2016, Up to 02 months
Population: RS
Measure: Number; unit: Percentage of participants
Arm/Group | Nintedanib Plus Capecitabine
Number analyzed (Participants) | 1
Percentage of participants | NA — Since only one patient was enrolled prior to termination of the trial, no data summarization or analysis was carried out.

5. Secondary Outcome: Percentage of Patients With Grade 3 or Worse Adverse Events
Description: Percentage of patients with grade 3 or worse adverse events.
Time Frame: Data collected up to cut-off date 09 Sep 2016, Up to 02 months
Population: RS
Measure: Number; unit: Percentage of participants
Arm/Group | Nintedanib Plus Capecitabine
Number analyzed (Participants) | 1
Percentage of participants | 0

ADVERSE EVENTS:
Time Frame: From first drug administration till end of trial; up to 3 months
Arm/Group | Nintedanib Plus Capecitabine
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib Plus Capecitabine (N=1)
Decreased appetite (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 1

LIMITATIONS AND CAVEATS:
Trial was terminated prematurely because it was determined that nintedanib monotherapy demonstrated lack of efficacy in this indication in pivotal Phase III trial (LUME-Colon 1) that was ongoing at the time of the initiation of this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No